CLINICAL TRIAL: NCT06194513
Title: Examining the Effect of Oral Motor Intervention Applied to Preterm Babies by Their Mothers at Different Frequencies on Oral Feeding Performance and Mother Baby Bonding
Brief Title: Oral Motor Intervention to Preterms by Their Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2023.1690
Record Dates: First submitted 2023-12-20; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Premature
Keywords: The Motor to Infant Bonding Scale; Preterm Infant Oral Feeding Readiness Assessment; The Breastfeeding Assessment Tool
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The infants included in the study will be divided to 3 groups and will be treated at the same time as a control group and 2 treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1: Twice a day for 1 week PIOMI (Experimental): Mothers of preterm babies in this group who have oral feeding difficulties will be taught Oral Motor Intervention (PIOMI) and asked to apply it. During the applications, visual monitoring of the application will be provided via video call, and objective monitoring of the application will be provided with the PIOMI Reliability Assessment Tool.
  Interventions: Other: Intervention 1: Twice a day for 1 week PIOMI
- Intervention 2: Once a day for 2 weeks PIOMI (Experimental): Mothers of preterm babies in this group who have oral feeding difficulties will be taught Oral Motor Intervention (PIOMI) and asked to apply it. During the applications, visual monitoring of the application will be provided via video call, and objective monitoring of the application will be provided with the PIOMI Reliability Assessment Tool.
  Interventions: Other: Intervention 2: Once a day for 2 weeks PIOMI
- Control (No Intervention): In the control group, no extra intervention will be given to preterm babies who have difficulty in oral feeding, and oral activation will be provided only with a pacifier.

INTERVENTIONS:
Other: Intervention 1: Twice a day for 1 week PIOMI — Preterm babies will receive two sessions of treatment every day for a week, for a total of 14 sessions. Each session will be five minutes. The application is done at a time when the baby is peaceful and not very hungry. When the application is performed, the baby is positioned on his back and in a way that feels comfortable.
  Arms: Intervention 1: Twice a day for 1 week PIOMI
Other: Intervention 2: Once a day for 2 weeks PIOMI — Preterm babies will receive a total of 14 sessions of treatment, one every day for two weeks. Each session will be five minutes. The application is done at a time when the baby is peaceful and not very hungry. When the application is performed, the baby is positioned on his back and in a way that feels comfortable.
  Arms: Intervention 2: Once a day for 2 weeks PIOMI

SUMMARY:
Babies who have been discharged from the neonatal intensive care unit and have difficulty in oral feeding will be identified. Oral Motor Intervention (PIOMI) will be taught to the mothers of these babies and asked to practice. As a result of this application, the change in oral feeding skills in babies and its effect on mother-infant bonding will be evaluated.

DETAILED DESCRIPTION:
The aim of this study is to observe the changes in babies' oral feeding skills and mothers' mother-baby attachment evaluation status as a result of oral motor intervention (PIOMI) applied to preterms with oral feeding difficulties.

An estimated 20 million babies are born preterm (before the 37th week of gestation) each year in the world, and this number is increasing, and complications of prematurity are among the leading causes of death among children under 5 years of age. Three-quarters of these deaths are preventable with current, cost-effective interventions.

Problems experienced after discharge include delayed feeding ability, food rejection, difficulty in transitioning to solid foods, and slowdown in growth. The reasons that lead to these difficulties are; These are post-discharge health problems such as immaturity, parenteral or tube feeding as opposed to oral motor experience, and neurological or cognitive disorders. All of these make it difficult for the child to develop nutritional skills and cause stress, depression, and self-confidence in the family.

Premature Infant Oral Motor Intervention (PIOMI) is a five-minute, eight-step oral motor intervention applied to preterm infants that aims to mimic the in utero oral experience that strengthens and improves feeding mechanisms. PIOMI provides assisted movement to activate muscle contraction for suckling and oral feeding, generating force to move against resistance, increasing functional response to pressure. It improves control of movements in accordance with a specific protocol that includes light contact with fingertips on the lips, cheeks, chin, gums, palate and tongue for the first three minutes, and pacifier/thumb sucking for the last two minutes. It was developed by Lessen BS to provide oral motor stimulation in preterm babies and its reliability study was conducted. The Turkish adaptation of the application was made by Selver Güler and Zerrin Çiğdem in 2021.

This oral motor intervention will be taught to the mother by a physiotherapist trained in this field, and it is planned that the mother will perform the application. In this way, premature babies with low immunity will not risk their health and will be given the opportunity to be treated more safely at home rather than in a hospital environment, which will save time and money. The effect of oral motor intervention frequency on oral motor skills will also be examined through applications at different frequencies.

Before the applications and after all the applications are completed, LATCH (Breastfeeding Assessment Tool) and POFRAS (Oral Feeding Readiness Assessment Scale in Preterm Babies) are filled in by the physiotherapist to evaluate the oral motor skills of the babies, and ABBÖ (Mother Baby Attachment Scale) is filled in by the mother to observe the mother-baby attachment status.

Preterm (<37 weeks of gestation) and babies with a corrected age of up to 3 months will be evaluated. Medical records and demographic data of the babies, whose verbal and written consent has been obtained from their parents, will be collected and PIOMI will be applied to the babies in the intervention groups by their mothers at different frequencies (twice a day for 1 week, once a day for 2 weeks). In addition to these two groups, there will be a control group and the evaluation results of the 3 groups will be examined. It is planned to apply different frequencies to the babies in Groups 1 and 2. and Group 3/Control group will be given oral activation only with a pacifier for 14 days.

The sample size of this study was calculated using the G*Power 3.1.9.2 program. In the analysis, there was a medium effect size (f = 0.25), Type I α = 0.05 and 80% power, which should be included in each group. The number of participants was calculated as 42 people in total, 14 people per group.

With this thesis, the investigators aim to shed light on future studies by contributing to the literature and to observe the positive effect of this situation on both the baby and the mother by initiating an oral motor intervention in which the mother can directly participate in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the study is accepted by the family
* PIOMI can be applied and whose clinical condition is stable,
* Born earlier than 37 weeks,
* Those who have not been diagnosed with any disorder in swallowing functions,
* Without congenital anomalies and systemic diseases,
* Vital signs are stable,
* Babies without congenital anomalies or serious complications

Exclusion Criteria:

* Participation in the study is not accepted by their family,
* Those with congenital anomalies and systemic diseases.
* Those who have been diagnosed with swallowing disorder,
* Those with congenital disorders or birth trauma,
* Diagnosed with severe asphyxia,
* Those with intraventricular bleeding,
* Those with Neonatal Abstinence Syndrome,
* Those with Fetal Alcohol Syndrome,
* Babies connected to a ventilator

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
The LATCH Breastfeeding Assessment Tool (Latch Audible Swallowing, Type of Nipple, Comfort of Breast/Nipple, H-Hold/ Position) | 0, 7. day, 14. day
  LATCH is a tool created by analogy with the Apgar score system in terms of scoring method, and its evaluation is quick and easy.
  The Turkish validity of the Assessment Tool was conducted by Demirhan in 1997, Koyun in 2001, and Yenal and Okumuş in 2003, and it was recommended to be used as a reliable tool. The highest score that can be obtained from the scale is 10 and the lowest score is 0. Increasing scores from the scale indicate breastfeeding success. Cronbach Alpha value of the LATCH Breastfeeding Assessment Tool; Yenal and Okumuş found it as 0.95, Demirhan as 0.94, and Koyun as 0.96.
  The scale considers mother and baby together. It can be evaluated by a healthcare professional or the mother. In the evaluation; It includes the criteria for breast retention, the baby's swallowing movement, the type of nipple, the mother's comfort with the breast and nipple, and the position of holding the baby.
Preterm Infant Oral Feeding Readiness Assessment (PIOFRA/ POFRAS) | 0, 7. day, 14. day
  This scale consists of 5 categories (corrected gestational age, behavioral organization, mouth posture, oral reflexes, non-nutritive sucking) and 18 items and evaluates readiness for oral feeding in preterm infants. The scale is scored between 0-2 and the maximum score is 36. The cut-off point for switching a preterm baby to oral feeding was determined as 30 .
  Turkish Validity-Reliability: In the Turkish adaptation of this scale made by Çamur and Çetinkaya in 2020, the cut-off point was found to be 29.

SECONDARY OUTCOMES:
The Mother to Infant Bonding Scale (MIBS) | 0, 7. day, 14. day
  The scale is designed to be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word. This scale, which can be easily and quickly applied by the mother and father alone, shows the relationship between the bond established and the mother's early mood.
  MIBS is a 4-point Likert scale consisting of 8 items. Responses consisting of four options are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 24. In the evaluation, the 1st, 4th, and 6th items express positive emotions and are scored as 0, 1, 2, 3, while the 2nd, 3rd, 5th, 7th items are scored as 0, 1, 2, 3. Items 1 and 8 are expressions of negative emotions and are scored in reverse, as 3, 2, 1, 0.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Demirci, PT, Principal Investigator — Marmara University; Evrim Karadag Saygi, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegazy SM. Late Preterm Infants. A Guide for Nurses, Midwives, Clinicians, and Allied Health Professionals. Saudi Med J. 2019 Dec;40(12):1303. doi: 10.15537/smj.2019.12.24665. PMID 31828286
- [Background] Cerro N, Zeunert S, Simmer KN, Daniels LA. Eating behaviour of children 1.5-3.5 years born preterm: parents' perceptions. J Paediatr Child Health. 2002 Feb;38(1):72-8. doi: 10.1046/j.1440-1754.2002.00728.x. PMID 11869405
- [Background] Gewolb IH, Vice FL. Maturational changes in the rhythms, patterning, and coordination of respiration and swallow during feeding in preterm and term infants. Dev Med Child Neurol. 2006 Jul;48(7):589-94. doi: 10.1017/S001216220600123X. PMID 16780629
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525
- [Background] Fujinaga CI, de Moraes SA, Zamberlan-Amorim NE, Castral TC, de Almeida e Silva A, Scochi CG. Clinical validation of the Preterm Oral Feeding Readiness Assessment Scale. Rev Lat Am Enfermagem. 2013 Jan-Feb;21 Spec No:140-5. doi: 10.1590/s0104-11692013000700018. English, Portuguese. PMID 23459901